CLINICAL TRIAL: NCT03129009
Title: Changes of Hemodynamics and Vital Organ Function in Intracerebral Hemorrhage During Different General Anesthesia
Brief Title: Hemodynamics and Vital Organ Function in Intracerebral Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin Dong Liu, Principal Investigator, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XYFY-2017-008
Record Dates: First submitted 2017-03-29; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Balanced Anesthesia; Intracerebral Hemorrhage; Total Intravenous Anesthesia
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Balanced Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total intravenous anesthesia group (Active Comparator): Total intravenous anesthesia induced with sufentanil,etomidate,cisatracurium and midazolam and maintained with propofol,cisatracurium and remifentanil target controlled infusion
  Interventions: Drug: Total intravenous anesthesia group
- Balanced anesthesia group (Experimental): Balanced anesthesia induced with sufentanil,etomidate,cisatracurium and midazolam and maintained with cisatracurium and remifentanil target controlled infusion and sevoflurane inhalation
  Interventions: Drug: Balanced anesthesia group

INTERVENTIONS:
Drug: Total intravenous anesthesia group — Total intravenous anesthesia induced with sufentanil,etomidate,cisatracurium and midazolam and maintained with propofol,cisatracurium and remifentanil target controlled infusion
  Other Names: TIVA
  Arms: Total intravenous anesthesia group
Drug: Balanced anesthesia group — Balanced anesthesia induced with sufentanil,etomidate,cisatracurium and midazolam and maintained with cisatracurium and remifentanil target controlled infusion and sevoflurane inhalation
  Other Names: Balanced anesthesia
  Arms: Balanced anesthesia group

SUMMARY:
Spontaneous non-traumatic intracerebral hemorrhage (ICH) is a common symptom in clinical practice and is the most serious among all types of stroke.Recently, as a relatively mainstream and recognized INTERACT2 (five well-known international studies in the cerebrovascular field: IMS-III, MR RESCUE, SYNTHESIS EXPANSION, INTERACT2, CHANCE) studies have shown that in patients with standard systolic blood pressure Early intensive antihypertensive therapy does not increase the incidence of death or serious adverse events. The above studies confirm the safety and efficacy of early potent depression.In 2017, Anesthesiology published a META analysis of intraoperative hypotension and blood pressure versus baseline fluctuations. The final outcome showed that 20% of blood pressure in the study was similar to MAP <65 mmHg, regardless of the duration of the duration There will be postoperative myocardial and renal damage. Ischemia is a very important cause of organ damage. Myocardial injury is closely related to the level of mean arterial pressure, while ischemia and ischemic reperfusion injury are closely related to postoperative acute renal injury.There is no targeted guideline for ICH perioperative blood pressure management, especially intraoperative blood pressure management, and no previous studies have studied most of the studies involving ICH patients with conservative treatment, ICH patients with surgical treatment There are few reports on blood pressure control during surgery.

DETAILED DESCRIPTION:
The general anesthesia used in craniotomy, whether intravenous anesthesia or total intravenous anesthesia, have a certain degree of blood pressure and lead to a decline in blood pressure, the study aims to spontaneous cerebral hemorrhage this special And to observe the changes of hemodynamics and the changes of heart and kidney function in ICH, and to explore the relationship between the anesthesia and the blood of ICH. The range of volatility.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years to90 years.
2. acute stroke symptoms caused by initial spontaneous intracerebral hemorrhage as determined by CT or MRI Blood: the screen area: 30-50ml; cerebellum parts:> 10ml.
3. GCS score> 5 points

Exclusion Criteria:

1. ICH is caused by other factors (anticoagulation associated with cerebral hemorrhage, arteriovenous malformations, tumors)
2. intracerebral hematoma is thought to be associated with trauma (simple intracerebral hemorrhage)
3. there are surgical contraindications.
4. history of ischemic stroke
5. acute spontaneous intracerebral hemorrhage before the presence of dementia or limb dysfunction (paralysis or aphasia.
6. preoperative combined with chronic kidney disease (standard for glomerular filtration rate below 60 ml · min-1 · 1.73 m2 or received dialysis).
7. anesthesia time shorter than 60 min or lack of relevant basic information.
8. while there is interference with the experimental results or follow-up of the disease (tumor, severe cardiovascular disease).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
MAP changes relative to the changes before induction | Intraoperative
  MAP changes relative to the changes before induction; <20%, 20% -30%, 30% -40%,> 40%MAP changes relative to the changes before induction; <20%, 20% -30%, 30% -40%,> 40%

SECONDARY OUTCOMES:
All-cause mortality | 7 days post surgery
  All-cause mortality is the ratio of the total number of deaths resulting from a variety of causes over a period of time to the average population of the population over the same period.
Acute renal failure | 7 days post surgery
  Increased absolute serum creatinine ≥0.3mg / dl (≥26.5μmol / l), or ≥50% increase (1.5 times the baseline), or urine <0.5ml / (kg.h) for more than 6 hours Obstructive nephropathy or dehydration status)
CK-MB release level | 6 hour, 12 hour,24 hour,48 hour post surgery
  Clinically, CK-MB more than the total activity of CK 3 (ion exchange column chromatography) or 10 (immunosuppressive method) as the basis for the diagnosis of acute myocardial infarction.
Troponin T | 6 hour, 12 hour, 24 hour, 48 hour post surgery
  The levels of troponin T were released before anesthesia induction at 6 hour, 12 hour, 24 hour and 48 hour
Serum creatinine | 24 hour, 48 hour,72 hour post surgery
  Serum creatinine levels were measured before and after anesthesia induction at 24 hour, 48 hour

CONTACTS AND LOCATIONS:
Overall Officials: Jin Dong Liu, M.S, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available when this trial is finished and the article have been published

REFERENCES:
- [Result] Qureshi AI, Tuhrim S, Broderick JP, Batjer HH, Hondo H, Hanley DF. Spontaneous intracerebral hemorrhage. N Engl J Med. 2001 May 10;344(19):1450-60. doi: 10.1056/NEJM200105103441907. No abstract available. PMID 11346811
- [Result] Liu M, Wu B, Wang WZ, Lee LM, Zhang SH, Kong LZ. Stroke in China: epidemiology, prevention, and management strategies. Lancet Neurol. 2007 May;6(5):456-64. doi: 10.1016/S1474-4422(07)70004-2. PMID 17434100
- [Result] van Asch CJ, Luitse MJ, Rinkel GJ, van der Tweel I, Algra A, Klijn CJ. Incidence, case fatality, and functional outcome of intracerebral haemorrhage over time, according to age, sex, and ethnic origin: a systematic review and meta-analysis. Lancet Neurol. 2010 Feb;9(2):167-76. doi: 10.1016/S1474-4422(09)70340-0. Epub 2010 Jan 5. PMID 20056489
- [Result] Mayer SA, Rincon F. Treatment of intracerebral haemorrhage. Lancet Neurol. 2005 Oct;4(10):662-72. doi: 10.1016/S1474-4422(05)70195-2. PMID 16168935
- [Result] Mendelow AD, Gregson BA, Fernandes HM, Murray GD, Teasdale GM, Hope DT, Karimi A, Shaw MD, Barer DH; STICH investigators. Early surgery versus initial conservative treatment in patients with spontaneous supratentorial intracerebral haematomas in the International Surgical Trial in Intracerebral Haemorrhage (STICH): a randomised trial. Lancet. 2005 Jan 29-Feb 4;365(9457):387-97. doi: 10.1016/S0140-6736(05)17826-X. PMID 15680453
- [Result] Qureshi AI, Ezzeddine MA, Nasar A, Suri MF, Kirmani JF, Hussein HM, Divani AA, Reddi AS. Prevalence of elevated blood pressure in 563,704 adult patients with stroke presenting to the ED in the United States. Am J Emerg Med. 2007 Jan;25(1):32-8. doi: 10.1016/j.ajem.2006.07.008. PMID 17157679
- [Result] Zhang Y, Reilly KH, Tong W, Xu T, Chen J, Bazzano LA, Qiao D, Ju Z, Chen CS, He J. Blood pressure and clinical outcome among patients with acute stroke in Inner Mongolia, China. J Hypertens. 2008 Jul;26(7):1446-52. doi: 10.1097/HJH.0b013e328300a24a. PMID 18551022
- [Result] Rodriguez-Luna D, Pineiro S, Rubiera M, Ribo M, Coscojuela P, Pagola J, Flores A, Muchada M, Ibarra B, Meler P, Sanjuan E, Hernandez-Guillamon M, Alvarez-Sabin J, Montaner J, Molina CA. Impact of blood pressure changes and course on hematoma growth in acute intracerebral hemorrhage. Eur J Neurol. 2013 Sep;20(9):1277-83. doi: 10.1111/ene.12180. Epub 2013 May 5. PMID 23647568
- [Result] Sakamoto Y, Koga M, Yamagami H, Okuda S, Okada Y, Kimura K, Shiokawa Y, Nakagawara J, Furui E, Hasegawa Y, Kario K, Arihiro S, Sato S, Kobayashi J, Tanaka E, Nagatsuka K, Minematsu K, Toyoda K; SAMURAI Study Investigators. Systolic blood pressure after intravenous antihypertensive treatment and clinical outcomes in hyperacute intracerebral hemorrhage: the stroke acute management with urgent risk-factor assessment and improvement-intracerebral hemorrhage study. Stroke. 2013 Jul;44(7):1846-51. doi: 10.1161/STROKEAHA.113.001212. Epub 2013 May 23. PMID 23704107
- [Result] Butcher KS, Jeerakathil T, Hill M, Demchuk AM, Dowlatshahi D, Coutts SB, Gould B, McCourt R, Asdaghi N, Findlay JM, Emery D, Shuaib A; ICH ADAPT Investigators. The Intracerebral Hemorrhage Acutely Decreasing Arterial Pressure Trial. Stroke. 2013 Mar;44(3):620-6. doi: 10.1161/STROKEAHA.111.000188. Epub 2013 Feb 7. PMID 23391776
- [Result] Arima H, Huang Y, Wang JG, Heeley E, Delcourt C, Parsons M, Li Q, Neal B, Chalmers J, Anderson C; INTERACT1 Investigators. Earlier blood pressure-lowering and greater attenuation of hematoma growth in acute intracerebral hemorrhage: INTERACT pilot phase. Stroke. 2012 Aug;43(8):2236-8. doi: 10.1161/STROKEAHA.112.651422. Epub 2012 Jun 7. PMID 22678090
- [Result] Arima H, Anderson CS, Wang JG, Huang Y, Heeley E, Neal B, Woodward M, Skulina C, Parsons MW, Peng B, Tao QL, Li YC, Jiang JD, Tai LW, Zhang JL, Xu E, Cheng Y, Morgenstern LB, Chalmers J; Intensive Blood Pressure Reduction in Acute Cerebral Haemorrhage Trial Investigators. Lower treatment blood pressure is associated with greatest reduction in hematoma growth after acute intracerebral hemorrhage. Hypertension. 2010 Nov;56(5):852-8. doi: 10.1161/HYPERTENSIONAHA.110.154328. Epub 2010 Sep 7. PMID 20823381
- [Result] Anderson CS, Heeley E, Huang Y, Wang J, Stapf C, Delcourt C, Lindley R, Robinson T, Lavados P, Neal B, Hata J, Arima H, Parsons M, Li Y, Wang J, Heritier S, Li Q, Woodward M, Simes RJ, Davis SM, Chalmers J; INTERACT2 Investigators. Rapid blood-pressure lowering in patients with acute intracerebral hemorrhage. N Engl J Med. 2013 Jun 20;368(25):2355-65. doi: 10.1056/NEJMoa1214609. Epub 2013 May 29. PMID 23713578
- [Result] Zheng J, Lin S, Li H, Ma J, Guo R, Fang Y, Ma L, Liu W, Liu M, You C. Perioperative antihypertensive treatment in patients of spontaneous intracerebral hemorrhage (PATICH): a clinical trial protocol. Contemp Clin Trials. 2014 Sep;39(1):9-13. doi: 10.1016/j.cct.2014.06.015. Epub 2014 Jul 2. PMID 24999076
- [Result] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Result] POISE Study Group; Devereaux PJ, Yang H, Yusuf S, Guyatt G, Leslie K, Villar JC, Xavier D, Chrolavicius S, Greenspan L, Pogue J, Pais P, Liu L, Xu S, Malaga G, Avezum A, Chan M, Montori VM, Jacka M, Choi P. Effects of extended-release metoprolol succinate in patients undergoing non-cardiac surgery (POISE trial): a randomised controlled trial. Lancet. 2008 May 31;371(9627):1839-47. doi: 10.1016/S0140-6736(08)60601-7. Epub 2008 May 12. PMID 18479744
- [Result] Lienhart A, Auroy Y, Pequignot F, Benhamou D, Warszawski J, Bovet M, Jougla E. Survey of anesthesia-related mortality in France. Anesthesiology. 2006 Dec;105(6):1087-97. doi: 10.1097/00000542-200612000-00008. PMID 17122571
- [Result] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Result] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Result] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768
- [Result] Liu JD, Chen HJ, Wang DL, Wang H, Deng Q. Pim-1 Kinase Regulating Dynamics Related Protein 1 Mediates Sevoflurane Postconditioning-induced Cardioprotection. Chin Med J (Engl). 2017 Feb 5;130(3):309-317. doi: 10.4103/0366-6999.198922. PMID 28139514
- [Result] Yang L, Xie P, Wu J, Yu J, Yu T, Wang H, Wang J, Xia Z, Zheng H. Sevoflurane postconditioning improves myocardial mitochondrial respiratory function and reduces myocardial ischemia-reperfusion injury by up-regulating HIF-1. Am J Transl Res. 2016 Oct 15;8(10):4415-4424. eCollection 2016. PMID 27830025
- [Result] Runzer TD, Ansley DM, Godin DV, Chambers GK. Tissue antioxidant capacity during anesthesia: propofol enhances in vivo red cell and tissue antioxidant capacity in a rat model. Anesth Analg. 2002 Jan;94(1):89-93, table of contents. doi: 10.1097/00000539-200201000-00017. PMID 11772807
- [Result] Xia Z, Godin DV, Chang TK, Ansley DM. Dose-dependent protection of cardiac function by propofol during ischemia and early reperfusion in rats: effects on 15-F2t-isoprostane formation. Can J Physiol Pharmacol. 2003 Jan;81(1):14-21. doi: 10.1139/y02-170. PMID 12665253
- [Result] Xia Z, Godin DV, Ansley DM. Propofol enhances ischemic tolerance of middle-aged rat hearts: effects on 15-F(2t)-isoprostane formation and tissue antioxidant capacity. Cardiovasc Res. 2003 Jul 1;59(1):113-21. doi: 10.1016/s0008-6363(03)00351-1. PMID 12829182
- [Result] Wang B, Shravah J, Luo H, Raedschelders K, Chen DD, Ansley DM. Propofol protects against hydrogen peroxide-induced injury in cardiac H9c2 cells via Akt activation and Bcl-2 up-regulation. Biochem Biophys Res Commun. 2009 Nov 6;389(1):105-11. doi: 10.1016/j.bbrc.2009.08.097. Epub 2009 Aug 22. PMID 19703415